CLINICAL TRIAL: NCT02237053
Title: A Prospective Randomized, Placebo (Saline)-Controlled, Balanced, 3-treatment Regimen Crossover Study Comparing the Effects of Prolonged (13 h) Hyperglucagonemia With Those of Acute (3 hr) Hyperglucagonemia on Energy Expenditure and Endogenous Glucose Protection (EGP).
Brief Title: Effects of Glucagon Administration on Energy Expenditure
Acronym: GLEE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TRIMDFH 601205
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hyperglucagonemia; Obesity
Keywords: Energy expenditure; Glucagon; Octreotide; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Glucagon; Octreotide; Sodium Chloride; Insulin; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glucagon with Octreotide and insulin (Active Comparator): Overnight (10 hours) infusion of glucagon, then 3 hours infusion of glucagon with concurrent infusions of Octreotide and insulin.
  Interventions: Drug: Glucagon; Drug: Octreotide; Drug: Insulin
- Placebo, Glucagon with Octreotide and Insulin (Placebo Comparator): Overnight (10 hours) infusion of saline, then 3 hour infusion of glucagon with concurrent infusions of Octreotide and insulin.
  Interventions: Drug: Glucagon; Drug: Octreotide; Behavioral: Placebo; Drug: Insulin
- Placebo, with Octreotide and insulin (Placebo Comparator): Overnight (10 hours) infusion of saline, then 3 hour infusion of saline with concurrent infusions of Octreotide and insulin.
  Interventions: Drug: Octreotide; Behavioral: Placebo; Drug: Insulin

INTERVENTIONS:
Drug: Glucagon
  Arms: Glucagon with Octreotide and insulin; Placebo, Glucagon with Octreotide and Insulin
Drug: Octreotide
  Other Names: Sandostatin
Behavioral: Placebo
  Other Names: Saline
  Arms: Placebo, Glucagon with Octreotide and Insulin; Placebo, with Octreotide and insulin
Drug: Insulin
  Other Names: Hypoglycemic agent

SUMMARY:
The purpose of this study is to collect data to help researchers better understand the effects of glucagon on the amount of calories burned.

DETAILED DESCRIPTION:
1. To compare the effect of prolonged hyperglucagonemia to that of acute hyperglucagonemia on energy expenditure in healthy subjects using room indirect calorimetry in the setting of octreotide-mediated prevention of plasma insulin excursions.
2. To compare the effects of prolonged hyperglucagonemia to acute hyperglucagonemia on EGP in healthy subjects in the setting of octreotide-mediated prevention of plasma insulin excursions.
3. To determine the effects of prolonged hyperglucagonemia to acute hyperglucagonemia on rates of substrate oxidation, fibroblast growth factor21 and metabolites of interest.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male between the ages of 18 and 50 years.
* Subject has a body mass index (BMI) less than or equal to 26 kg/m2. BMI = weight (kg)/height (m) and body weight greater than or equal to 50 kg at the pre-study (screening) visit
* Subject has been weight stable over the last 3 months (plus or minus 3 kg)
* Subject is judged to be non-diabetic and in good health on the basis of medical history, physical examination, electrocardiogram, and routine laboratory data.
* Subject understands the procedures and agrees to participate in the study program by giving written informed consent, and is willing to comply with the trial restrictions.
* Subject is willing to avoid alcohol consumption for 48 hours prior to each period.
* Subject is willing to avoid strenuous physical activity (i.e., strenuous or unaccustomed weight lifting, running, bicycling, etc.) beginning 72 hours prior to first drug administration period and for the duration of the study.
* Subject is willing to avoid consumption of caffeine and caffeinated beverages for 24 hours prior to drug administration in each period. Subject is willing to consume no more than 2 caffeinated beverages per day during all other parts of the study.

Exclusion Criteria:

* is mentally or legally incapacitated, has significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years. Subjects who have had situational depression may be enrolled in the trial at the discretion of the investigator.
* has a history of clinically significant endocrine (including type 1 or type 2, or steroid-induced diabetes), gastrointestinal (including prior history of pancreatitis), cardiovascular (including hypertension, angina, coronary artery disease, valvular disease, heart rate or rhythm abnormalities), hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases. Subjects with a history of uncomplicated kidney stones or childhood asthma may be enrolled in the trial at the discretion of the investigator.
* has a known history of any endocrine tumors (e.g. pheochromocytoma, glucagonoma, or insulinoma, etc.)
* has a clinically significant abnormality on screening ECG or evidence or a history of myocardial ischemia, atrioventricular block, Wolf-Parkinson-White syndrome or other conduction abnormality. Subjects having any clinically significant ECG abnormality at screening may be included at the discretion of the PI.
* has a fasting blood glucose (FPG) less than or equal to 65 mg/dL or greater than or equal to 100 mg/dL on the pre-study screening labs.
* has impaired kidney or liver function, as evidenced by screening blood work.
* has irritable bowel disease, or recurrent occurrences of nausea, vomiting, diarrhea, constipation or abdominal pain.
* has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* has an estimated creatinine clearance of ≤80 mL/min based on the Cockcroft-Gault equation
* has a history of neoplastic disease
* has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food; or allergy/intolerability to insulin, glucagon, or octreotide.
* is positive for hepatitis B surface antigen, hepatitis C antibodies, or HIV
* had major surgery within 3 months, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* has participated in another investigational trial within 4 weeks prior to the pretrial (screening) visit. The 4 week window will be derived from the date of the last trial medication and / or blood collection in a previous trial and/or adverse event related to trial drug to the pretrial/screening visit of the current trial.
* consumes greater than 2 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day. Patients that consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* consumes excessive amounts, defined as greater than 4 servings

  (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day.
* is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months of the screening visit.
* is unwilling or unable to adhere to the dietary needs during the study, or to consume the standardized meals during the study, and/or is on a carbohydrate restricted diet (i.e., a diet <100 grams per day of carbohydrate).
* is any concern by the investigator regarding the safe participation of the subject in the trial or for any other reason; the investigator considers the subject inappropriate for participation in the trial.
* has a history of claustrophobia or is claustrophobic.
* has ever had an organ transplant.
* is a smoker or uses other nicotine-containing products (for at least 6 months prior to drug administration); plans to begin smoking or using nicotine-containing products during the conduct of the study.
* has poor intravenous access.
* has used any medications that are known to influence glucose, fat, or energy metabolism within the last 3 months (growth hormones, steroids, etc.)
* has blood pressure at screening visit less than or equal to 100/50 mm Hg or greater than or equal to 160/100 mm Hg.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measure of energy expenditure | Day 2, Day 9, Day 16
  Energy expenditure (and respiratory quotient) will be measured within the small calorimeter rooms. Oxygen and carbon dioxide levels in the chambers will be measured.

SECONDARY OUTCOMES:
Measure of endogenous glucose production | Day 3, Day 10, Day 17
  The measure of endogenous glucose production will be calculated from the deuterated glucose infusion rate and the plasma deuterated glucose enrichment using the non-steady state equation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Florida Hospital Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Flint A, Raben A, Rehfeld JF, Holst JJ, Astrup A. The effect of glucagon-like peptide-1 on energy expenditure and substrate metabolism in humans. Int J Obes Relat Metab Disord. 2000 Mar;24(3):288-98. doi: 10.1038/sj.ijo.0801126. PMID 10757621
- [Background] Cryer PE. Minireview: Glucagon in the pathogenesis of hypoglycemia and hyperglycemia in diabetes. Endocrinology. 2012 Mar;153(3):1039-48. doi: 10.1210/en.2011-1499. Epub 2011 Dec 13. PMID 22166985
- [Background] SCHULMAN JL, CARLETON JL, WHITNEY G, WHITEHORN JC. Effect of glucagon on food intake and body weight in man. J Appl Physiol. 1957 Nov;11(3):419-21. doi: 10.1152/jappl.1957.11.3.419. No abstract available. PMID 13480952
- [Background] Nair KS. Hyperglucagonemia increases resting metabolic rate in man during insulin deficiency. J Clin Endocrinol Metab. 1987 May;64(5):896-901. doi: 10.1210/jcem-64-5-896. PMID 2881943
- [Background] Calles-Escandon J. Insulin dissociates hepatic glucose cycling and glucagon-induced thermogenesis in man. Metabolism. 1994 Aug;43(8):1000-5. doi: 10.1016/0026-0495(94)90180-5. PMID 8052138
- [Background] Miyoshi H, Shulman GI, Peters EJ, Wolfe MH, Elahi D, Wolfe RR. Hormonal control of substrate cycling in humans. J Clin Invest. 1988 May;81(5):1545-55. doi: 10.1172/JCI113487. PMID 3284915
- [Background] Billington CJ, Briggs JE, Link JG, Levine AS. Glucagon in physiological concentrations stimulates brown fat thermogenesis in vivo. Am J Physiol. 1991 Aug;261(2 Pt 2):R501-7. doi: 10.1152/ajpregu.1991.261.2.R501. PMID 1877708
- [Background] Gimeno RE, Moller DE. FGF21-based pharmacotherapy--potential utility for metabolic disorders. Trends Endocrinol Metab. 2014 Jun;25(6):303-11. doi: 10.1016/j.tem.2014.03.001. Epub 2014 Apr 5. PMID 24709036
- [Background] Boyle PJ, Justice K, Krentz AJ, Nagy RJ, Schade DS. Octreotide reverses hyperinsulinemia and prevents hypoglycemia induced by sulfonylurea overdoses. J Clin Endocrinol Metab. 1993 Mar;76(3):752-6. doi: 10.1210/jcem.76.3.8445035.
- [Background] Krentz AJ, Boyle PJ, Macdonald LM, Schade DS. Octreotide: a long-acting inhibitor of endogenous hormone secretion for human metabolic investigations. Metabolism. 1994 Jan;43(1):24-31. doi: 10.1016/0026-0495(94)90153-8. PMID 8289671
- [Background] Tan TM, Field BC, McCullough KA, Troke RC, Chambers ES, Salem V, Gonzalez Maffe J, Baynes KC, De Silva A, Viardot A, Alsafi A, Frost GS, Ghatei MA, Bloom SR. Coadministration of glucagon-like peptide-1 during glucagon infusion in humans results in increased energy expenditure and amelioration of hyperglycemia. Diabetes. 2013 Apr;62(4):1131-8. doi: 10.2337/db12-0797. Epub 2012 Dec 17. PMID 23248172
- [Background] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org